CLINICAL TRIAL: NCT07207369
Title: A Multicenter, Cohort-design, Double-blind, Randomized, Parallel-group, Controlled Study to Evaluate the Safety and Effectiveness of ELAPR002f Injectable Gel in Adult Participants With Atrophic Acne Scars
Brief Title: A Study to Assess the Safety and Effectiveness of ELAPR002f Injectable Gel in Adult Participants With Atrophic Acne Scars
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-701-008
Record Dates: First submitted 2025-10-02; First posted 2025-10-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acne Scars
Keywords: Acne Scars; ELAPR002f injectable gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Cohort 1: Open-Label ELAPR002f Injectable Gel (Experimental): Participants will receive ELAPR002f Injectable Gel on Days 1, 31, and 61. Participants will be followed for up to 420 days.
  Interventions: Device: ELAPR002f Injectable Gel
- Cohort 2: ELAPR002f Injectable Gel (Experimental): Participants will receive ELAPR002f Injectable Gel on Days 1, 31, and 61. Participants will be followed for up to 420 days.
  Interventions: Device: ELAPR002f Injectable Gel
- Cohort 2: Saline Control (Experimental): Participants will receive a saline control on Days 1, 31, and 61. Participants will be followed for up to 420 days.
  Interventions: Device: Saline Control

INTERVENTIONS:
Device: ELAPR002f Injectable Gel — Intradermal Injections
  Arms: Cohort 1: Open-Label ELAPR002f Injectable Gel; Cohort 2: ELAPR002f Injectable Gel
Device: Saline Control — Intradermal Injections
  Arms: Cohort 2: Saline Control

SUMMARY:
Atrophic acne scars are flat, indented or with an inverted center scars that develop at the endpoint of the normal healing process for acne. Acne scarring that remains after acne resolves has a significant impact on health related quality of life, including reduced self-esteem and embarrassment/self consciousness. ELAPR002f provides an immediate space-occupying effect for filling in the scar tissue. The purpose of this study is to assess how safe and effective ELAPR002f injectable gel is on adult participants with atrophic acne scars.

ELAPR002f injectable gel is an investigational device being developed for the treatment of facial atrophic acne scars. There are 2 cohorts in this study. In Cohort 1, all participants will receive ELAPR002f injectable gel. In Cohort 2, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to the saline active control group. Around 395 adult participants with moderate to severe atrophic acne scarring on both cheeks will be screened in the study in approximately 25 sites in the United States.

Participants will receive 3 treatments over 2 months of intradermal injections of either ELAPR002f injectable gel or saline active control and will be followed for up to an additional 12 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health, and seeking improvement of atrophic acne scars.
* Moderate to severe atrophic acne scarring (Grade 4 or 5 on the Allergan Acne Scar Improvement Scale [ASIS]) on each cheek based on evaluating investigator (EI) live assessment (both cheeks must qualify but do not need to have the same score) at the first Screening Visit.
* At least 5 rolling or boxcar-type acne scars in total within the predefined 4 cm × 4 cm assessment field of either cheek in areas of otherwise normal healthy skin, as assessed by the treating investigator (TI).

Exclusion Criteria:

* The participant has clinically significant acne on the face.
* Current cutaneous or mucosal inflammatory or infectious processes other than acne (eg, herpes), rosacea, abscess, an unhealed wound, or a cancerous or precancerous lesion, on the face.
* The participant presents with predominantly ice pick scars.
* History of keloid scar formation, hypertrophic scarring, and/or post inflammatory hyperpigmentation or hypopigmentation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a 20% Reduction in Acne Scar Area | Baseline to Day 181
  The acne scar area is calculated from 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the treating investigator (TI).
Number of Participants with Adverse Events | Up to Day 420
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Presence of Binding Antibodies | Up to Day 420
  Presence of binding antibodies followed by characterization through isotyping and evaluation of cross-reactivity to endogenous tissues.
Number of Participants with Injection Site Responses (ISRs) and Systemic Responses | Up to Day 420
  Incidence of ISRs/systemic responses as recorded by e-diary. ISRs are defined as redness, pain after injection, tenderness to touch, firmness, swelling, lumps/bumps, bruising, itching and discoloration (not redness or bruising).
Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Parameters | Up to Day 420
  Vital sign parameters include body temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters | Up to Day 420
  Clinical laboratory parameters include tests of hematology, chemistry, and urinalysis. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Physical Measurements | Up to Day 420
  Physical measurements include weight and BMI. The investigator will assess the results for clinical significance.
Change from Baseline Procedure Pain | Up to Day 420
  Participants will assess procedure pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) after each of the 3 treatment sessions.
Number of Participants with a Positive Skin Test | Up to Day 420
  Participants will undergo a skin test in the volar area of the forearm to test for hypersensitivity.
Number of Participants with Visual Disturbance Symptoms Associated with Vascular Occlusion | Up to Day 420
  Number of participants with any acute cognitive changes or any change in confrontational visual fields, ocular motility, or a worsening (1-line change or more) on the Snellen visual acuity assessment.
Number of Participants Needing a Histology of Volar Forearm Site Biopsy | Up to Day 420
  Participants who are suspected of having a hypersensitivity reaction or have a hypersensitivity reaction to the volar forearm injection site will require a punch biopsy of the volar forearm injection site.

SECONDARY OUTCOMES:
Change from Baseline on the Overall Score of ACNE-Q Acne Scars Questionnaire | Up to Day 420
  The ACNE-Q Acne Scars questionnaire includes 10 questions that ask how much the participant is bothered by their acne scars on a 4-point scale ranging from 1=Not at all to 4=Very Much.
Change from Baseline on the Overall Score of ACNE-Q - Appearance-Related Distress | Up to Day 420
  ACNE-Q - Appearance-Related Distress questionnaire includes 8 questions that ask about how the participants describe themselves on a 4-point scale ranging from 1=Never to 4=Always.
Change from Baseline on the Overall Score of FACE-Q Satisfaction with Skin Total Score | Up to Day 420
  FACE-Q Satisfaction With Skin questionnaire includes 12 questions that ask how much the participants are satisfied or dissatisfied with their facial skin on a 4-point scale ranging from 1=Very Dissatisfied to 4=Very Satisfied.
Percentage of Participants Achieving "Responder" Status on Either Cheek Based on the Allergan Acne Scar Improvement Scale (ASIS), as assessed by the Evaluating Investigator | Up to Day 420
  A "responder" is a participant who achieves 1-grade improvement on either cheek based on the ASIS, as assessed by the EI. The ASIS is a 5-grade scale used to assess acne scar improvement ranging from 1=Almost None to 5=Severe. Each side of the face is scored separately.
Percentage of Participants who Achieve a 20% Reduction in Acne Scar Area | Up to Day 420
  The acne scar area is calculated from 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the treating investigator (TI).
Percent Change from Baseline in Acne Scar Area | Up to Day 420
  The acne scar area is measured by 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the TI.
Percent Change from Baseline in Acne Scar Volume | Up to Day 420
  The acne scar volume is measured by 3D camera imaging software. Volume is defined as the sum of the individual scar volume of the 5 most prominent scars identified by the TI.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - Advanced Research Associates - Glendale /ID# 254961, Glendale, Arizona
  - Marcus Facial Plastic Surgery /ID# 275880, Redondo Beach, California
  - Pacific Clinical Innovations /ID# 256185, Vista, California
  - DMR Research PLLC /ID# 256199, Westport, Connecticut
  - Hamilton Research, LLC /ID# 256925, Alpharetta, Georgia
  - Aesthetic Center at Woodholme /ID# 256197, Baltimore, Maryland
  - The Center for Dermatology Cosmetics & Laser Surgery /ID# 256182, Mount Kisco, New York
  - Wilmington Dermatology Center /ID# 256192, Wilmington, North Carolina
  - Austin Institute for Clinical Research - Pflugerville /ID# 256200, Pflugerville, Texas
  - SkinDC /ID# 254962, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=2015-701-008